CLINICAL TRIAL: NCT00903591
Title: Genome-Wide Association Study of Radiation Exposure and Bilateral Breast Cancer
Brief Title: Study of Radiation Exposure and Bilateral Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Translational Genomics Research Institute (Other); University of Southern California (Other); University of Virginia (Other); Lund University (Other); Ontario Cancer Registry (OCR) and Mount Sinai Hospital- Toronto (MSHT) (Unknown); Northern California Cancer Center (Other); Fred Hutchinson Cancer Center (Other); University of Iowa (Other); Danish Cancer Society (Other); Beckman Research Institute (Other); City of Hope National Medical Center (Other); M.D. Anderson Cancer Center (Other); Vanderbilt University School of Medicine (Other); NYU Langone Health (Other); University of Chicago (Other); University of California, Irvine (Other); Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 09-040; R01CA129639-01A2 (NIH)
Record Dates: First submitted 2009-05-15; First posted 2009-05-18 (Estimated); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Breast; cancer; 09-040; blood sample; saliva sample; WECARE; GWA
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Blood Specimen Collection; Cycloserine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample or saliva sample

GROUPS / COHORTS (1):
- 1: All women will be interviewed by telephone using the a similar questionnaire as used in the parent study. DNA samples will be obtained either via blood samples drawn during a home or clinic visits, or an Oragene Saliva DNA Self-Collection Kit sent to the participant's home.
  Interventions: Other: questionaire, blood or saliva sample

INTERVENTIONS:
Other: questionaire, blood or saliva sample — Take part in an approximately 45 minute telephone interview, with questions about detailed treatment (chemotherapy, hormonal therapy, radiation therapy (RT)) for all study participants. Their medical records will be reviewed to get further details about treatment of their breast cancer. They donate either a 35 ml blood sample (about 3 tablespoons) or a saliva sample. Blood Sample: if patient consents to give a blood sample, following the interview, they will be contacted by our staff phlebotomist (a person trained to draw blood). A scheduled appointment to draw a blood sample from you at your home. At the time of the blood draw, the phlebotomist will collect approximately 2 and 1/3 tablespoons of blood. Saliva Sample: if they choose not to give a blood sample, but consent to give a saliva sample instead, a saliva kit will be sent to there home. Once they provide the sample in the kit, they will be asked to mail back the sample in the pre-labeled kit that was sent to them.
  Other Names: The women who consented to 'future contact' in the WECARE:GWAS Study will be; identified, approached, and interviewed by investigative teams in the five data collection sites; (CPIC, MSHT, FHCRC, Iowa, and DCS) over approximately 8 months. Across all data; collection sites, we will approach all eligible cases and controls who consented to future contact; and request participation in the follow-up study to complete the structured questionnaire either; via mail or telephone.

SUMMARY:
This study is being done to find out what factors may be related to the risk of getting a second breast cancer among women who already have breast cancer in one breast. It will look at how genes, treatment for breast cancer; including radiation therapy, and the effects of different lifestyle activities, may affect the risk of breast cancer. It will use different processes to find genes that might increase the risk of breast cancer. The results of this study may help to develop better ways to detect, treat and prevent breast cancer. This study will compare women who have breast cancer in both breasts to women who have breast cancer in only one breast.

DETAILED DESCRIPTION:
This study expands upon an existing case-control study we call the Women's Environment Cancer and Radiation Epidemiology (WECARE) Study. For simplicity, in this protocol, we will refer to that study as the "parent" study. The goal of both studies is to examine the interaction of radiation exposure and genetic susceptibility factors in the etiology of breast cancer. A subset of study participants who consented to 'future contact' in the GWA Study (and those in the 'parent' study from selected sites) will be included in an analysis of radiation-related heart disease and related conditions.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for Cases: All women who meet the following eligibility requirements will be recruited as cases for the WECARE:GWA Study if they are not already cases (or refusers) from the parent WECARE Study:
* Diagnosed since 1/1/1990 with a histologically confirmed first primary breast cancer (only invasive stage 1 or 2) while residing in one of the study enrollment site (cancer registry);
* Diagnosed since 1/1/1992 with CBC (invasive only any stage) while residing in the same enrollment site (cancer registry);
* Two years or longer time interval between first and second primaries; Between the ages of 18 and 54 at the time of diagnosis of the first primary;
* Alive at time of contact; and
* No history of previous or intervening cancer diagnosis, except cervical cancer in situ (CIS) or non-melanoma skin cancer.
* Without bilateral mastectomy or prophylactic mastectomy of the contralateral breast following diagnosis of their first primary.

Eligibility for Controls: Women who meet all of the following requirements will be eligible as controls. One matched control will be recruited for each participating case:

* Diagnosed since 1/1/1990 with their first primary breast cancer (only invasive stage 1 or 2) while residing in one of the study enrollment site (i.e., cancer registry);
* Between the ages of 18 and 54 at the time of diagnosis of the first primary;
* Residing in the same study enrollment site (cancer registry) as when they were diagnosed with their breast cancer;
* Alive at time of contact;
* Never diagnosed (at reference date (date of first diagnosis plus "at risk interval" of matched case)) as having had CBC or any other cancer diagnosis other than the original breast cancer; with the exception of CIS or non-melanoma skin cancer.
* Without bilateral mastectomy or prophylactic mastectomy of the contralateral breast following diagnosis of their first primary.

Matching of Controls: Controls eligible for inclusion in this study will be individually matched (1:1) to cases on:

* Enrollment site (cancer registry);
* Age at diagnosis of the cases first primary(within 5-year age groups);
* Year of diagnosis of the cases first primary;(within 4-year categories);
* Race/ethnicity (white, black, Latina, Asian, other).

Exclusion Criteria:

Exclusion for Cases: Women with any of the following characteristics will be ineligible as a case:

* Unable to speak English in U.S. or Canadian enrolling sites or Spanish in the California site, and Danish in Denmark
* Unable to sign informed consent
* Stage IV distant metastases for either the first or second primary (lymph node metastasis is acceptable, but there should be no organ involvement
* Simultaneous diagnosis of invasive in one breast and in situ in the other breast

Exclusion for Controls: Women with any of the following characteristics will be ineligible as a control:

* Unable to speak English in U.S. and Canadian enrolling sites, or Spanish in the California site and Danish in Demark
* Unable to sign informed consent
* Stage IV distant metastases (lymph node metastasis is acceptable, but there should be no organ involvement

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All of the WECARE:GWA Study participants (new cases and individually matched controls) will be identified, recruited, and interviewed by investigative teams in the five population-based cancer registries (NCC, OCR, FHCRC, Iowa, and DCS).
Sampling Method: Non-Probability Sample
Enrollment: 1699 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Identify single nucleotide polymorphism's that are associated with contralateral breast cancer using a two-stage approach in a population-based case-control study. | 2.5 years

SECONDARY OUTCOMES:
Identify single nucleotide polymorphism that interact with radiation exposure. | 2.5 years
Replication. Using the entire WECARE Study population, determine whether genomic regions found to be associated with unilateral breast cancer as identified via independent genome-wide association studies conducted by other research groups. | 2.5 years
Characterize genomic regions containing variants associated with contralateral breast cancer and/or radiation-induced breast cancer in a population-based nested case-control study design. | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jonine Bernstein, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (4):
  - Stanford University, Stanford, California
  - University of Iowa, Iowa City, Iowa
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- ONTARIO CANCER REGISTRY, Mount Sinai Hospital, Toronto, Toronto, Ontario, Canada
- Danish Cancer Society, Copenhagen, Denmark

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org